CLINICAL TRIAL: NCT07049016
Title: Comparative Clinical Evaluation of Partial Coverage CAD/CAM Restoration Versus Nanohybrid Composite of Carious Hypomineralized Permanent Molars: A Randomized Controlled Trial
Brief Title: Comparing CAD/CAM vs Composite for Carious Hypomineralized Molars Evaluating Clinical Outcomes of Both Treatments.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Salmoon, Principal investigator, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-1
Record Dates: First submitted 2024-05-28; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct nanohybrid flowable composite (Active Comparator): is a bioactive flowable nano-hybrid restorative with a newly developed patented nanofiller. It is indicated for all classes including occlusal and cusp. It has all of the Giomer Technology attributes, anti-bacterial, acid neutralization, and fluoride release and recharge, with improved handling and effortless polishing, and maintains a long-lasting shine. Beautifil Flow Plus X has the strength, durability, and aesthetics of a hybrid composite
  Interventions: Other: restoring the MIH affected young permanent molars using Direct nanohybrid flowable composite
- IPS e.max CAD (Experimental): glass-ceramic-based restorations still offer the best translucency and esthetic qualities. The novel generation of lithium disilicate-based materials as IPS e.max CAD provides standard thickness and quick fabrication. Moreover, the adhesive technique used with this restoration type significantly raises its mechanical properties
  Interventions: Other: restoring the MIH affected young permanent molars using IPS e.max CAD

INTERVENTIONS:
Other: restoring the MIH affected young permanent molars using Direct nanohybrid flowable composite — (Shofu)is a bioactive flowable nano-hybrid restorative with a newly developed patented nanofiller. It is indicated for all classes including occlusal and cusp. It has all of the Giomer Technology attributes, anti-bacterial, acid neutralization, and fluoride release and recharge, with improved handling and effortless polishing, and maintains a long-lasting shine. Beautifil Flow Plus X has the strength, durability, and aesthetics of a hybrid composite.
  Arms: Direct nanohybrid flowable composite
Other: restoring the MIH affected young permanent molars using IPS e.max CAD — glass-ceramic-based restorations still offer the best translucency and esthetic qualities. The novel generation of lithium disilicate-based materials as IPS e.max CAD provides standard thickness and quick fabrication. Moreover, the adhesive technique used with this restoration type significantly raises its mechanical properties.
  Arms: IPS e.max CAD

SUMMARY:
Molar Incisor Hypomineralization (MIH) is enamel hypomineralization defined as qualitative defects caused by disruptions in either the calcification or maturation phases of amelogenesis affecting one or more first permanent molars (FPMs) and permanent incisors.

DETAILED DESCRIPTION:
Conventional treatment for such defects necessitates additional removal of the complete tooth structure to receive full crowns that cause more biologically harmful consequences like postoperative hypersensitivity and aggressive tooth structure loss. To fulfill the biological criteria for tooth preparation, conservatism is the major notion and goal that prosthodontists strive to achieve. Nowadays, minimally invasive techniques are frequently employed to support this idea. To meet the growing need for conservative and attractive tooth restorations, overlay ceramic restorations (covering all cusps) are becoming more necessary. These restorations show satisfactory mechanics, restoring function, and esthetic with preserving tooth structure Since all materials used to treat such cases, have distinct chemical compositions, they have different properties that affect their clinical outcome. Therefore, it is essential to compare them clinically because any restoration's clinical outcome affects its long-term success. According to the null hypothesis, different materials would not significantly affect the clinical result of ceramic overlay restorations.

Patients in all groups will receive a minimally invasive restoration with high esthetic advantages (Protection of the weak cusps and elimination of carious lesions with an esthetic way out) and long-term success of their MIH affected young permanent molars (either IPS e.max CAD, Direct nanohybrid flowable composite or VITA Suprinity PC-Glass ceramic (zirconia) that require minimal preparation depends on the type of restoration will receive.

ELIGIBILITY:
Inclusion Criteria:

1. 8-18 years old
2. Cooperative children with large carious First Permanent Molars (FPM) lesions associated with weak cusps and defected hypo-mineralized enamel.
3. Controlled dental disease - no active caries or periodontal diseases
4. Patients will be available to be clinically reviewed up to 1 year

Exclusion Criteria:

1. Patients with Symptoms of pulpitis.
2. Patients with uncontrolled active tooth decay or periodontal disease (i.e. 4+ mm probing depth and bleeding on probing).
3. Poor oral hygiene and motivation.
4. Patients with parafunctional habits (e.g., bruxism, biting on hard objects).
5. Patients with debilitating illnesses or complicating medical conditions

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Aesthetic Clinical success | 12 months (baseline ''1 day '', 6 and 12 months)
  According to FDI World Dental Federation criteria
  Five subcategories. From best to worst, the subcategories were:
  (1) clinically excellent, (2) clinically good, (3) clinically sufficient, (4) clinically not sufficient but repairable, and (5) clinically unacceptable. Assessment with category (5) was rated as a clinical failure.
Functional Clinical success | 12 months (baseline ''1 day '', 6 and 12 months)
  According to FDI World Dental Federation criteria
  Five subcategories. From best to worst, the subcategories were:
  (1) clinically excellent, (2) clinically good, (3) clinically sufficient, (4) clinically not sufficient but repairable, and (5) clinically unacceptable. Assessment with category (5) was rated as a clinical failure.
Biological clinical success | 12 months (baseline ''1 day '', 6 and 12 months)
  According to FDI World Dental Federation criteria
  Five subcategories. From best to worst, the subcategories were:
  (1) clinically excellent, (2) clinically good, (3) clinically sufficient, (4) clinically not sufficient but repairable, and (5) clinically unacceptable. Assessment with category (5) was rated as a clinical failure.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M. Attia, Ph.D, Principal Investigator — Lecturer of Fixed Prosthodontics MSA University
Locations (1):
- MSA University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT07049016/Prot_SAP_ICF_000.pdf